CLINICAL TRIAL: NCT00009776
Title: Combined Modality Radioimmunotherapy For Non-Hodgkin's Lymphoma With Three Cycles Of 90Y-DOTA-peptide-Lym-1, Paclitaxel and Cyclosporin A
Brief Title: Monoclonal Antibody Therapy, Paclitaxel, and Cyclosporine in Treating Patients With Recurrent or Refractory Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Davis (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068371; UCD-991869; NCI-V00-1641
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2001-10

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lym-1 monoclonal antibody; Cyclosporine; Paclitaxel; Indium

INTERVENTIONS:
Biological: monoclonal antibody Lym-1
Drug: cyclosporine
Drug: paclitaxel
Radiation: indium In 111 monoclonal antibody Lym-1
Radiation: yttrium Y 90 monoclonal antibody Lym-1

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining monoclonal antibody therapy with cyclosporine and paclitaxel may be an effective treatment for non-Hodgkin's lymphoma.

PURPOSE: Phase I trial to study the effectiveness of radiolabeled monoclonal antibody therapy combined with paclitaxel and cyclosporine in treating patients who have recurrent or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of yttrium Y 90 monoclonal antibody Lym-1 in combination with paclitaxel and cyclosporine in patients with recurrent or refractory non-Hodgkin's lymphoma.

OUTLINE: This is a dose-escalation study of yttrium Y 90 monoclonal antibody Lym-1 (Y90 MOAB Lym-1).

Patients receive oral cyclosporine every 12 hours on days -2 to 14. Patients receive unlabeled MOAB Lym-1 IV followed by a tracer dose of indium In 111 MOAB Lym-1 IV on day 0. On day 7, patients receive unlabeled MOAB Lym-1 IV followed by Y90 MOAB Lym-1 IV. Patients in cohorts 2-4 also receive paclitaxel IV over 3 hours on day 9. Courses repeat every 8 weeks for a total of 3 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3 patients receive escalating doses of Y90 MOAB Lym-1 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 patients experience dose-limiting toxicity.

Patients are followed monthly for 3 months, every 3 months for 21 months, and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study within 36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of non-Hodgkin's lymphoma (NHL) that has failed standard first-line chemotherapy
* Measurable disease
* NHL tissue Lym-1 reactive in vitro
* Normocellular bone marrow as evidenced by less than 25% of the bone marrow being NHL by bilateral bone marrow biopsy
* No bone marrow evidence of myelodysplastic syndrome
* HAMA titer negative

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* 3 to 6 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 130,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST no greater than 84 U/L

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* LVEF at least 50%

Pulmonary:

* FEV1 at least 60% of predicted
* FVC at least 60% of predicted
* DLCO at least 50%

Other:

* No other prior malignancy within the past 5 years except for nonmelanoma skin cancer
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior external beam radiotherapy

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-03

CONTACTS AND LOCATIONS:
Overall Officials: Gerald L. DeNardo, MD, Study Chair — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States